CLINICAL TRIAL: NCT03725098
Title: Prospective, Randomized, Controlled, Multicenter, Post-Market Clinical Study Evaluating the Performance of HEMOBLAST Bellows Compared to FLOSEAL Hemostatic Matrix in Cardiothoracic Operations
Brief Title: Clinical Study Evaluating the Performance of HEMOBLAST Bellows Compared to FLOSEAL Hemostatic Matrix in Cardiothoracic Operations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biom'Up France SAS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ETC 2018-005
Record Dates: First submitted 2018-10-08; First posted 2018-10-30 (Actual); Results first posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Cardiothoracic Surgery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- HEMOBLAST Bellows (Hemostatic Device) (Experimental): Bleeding sites will be treated with HEMOBLAST Bellows per its approved Indications for Use
  Interventions: Device: HEMOBLAST Bellows
- FLOSEAL (Hemostatic Device) (Active Comparator): Bleeding sites will be treated with FLOSEAL per its approved Indications for Use
  Interventions: Device: FLOSEAL

INTERVENTIONS:
Device: HEMOBLAST Bellows — The HEMOBLAST™ Bellows hemostatic agent consists of a bellows pre-loaded with 1.65g of powder composed of collagen, chondroitin sulfate, and thrombin (1500 IU). HEMOBLAST™ Bellows is indicated in surgical procedures as an adjunct to hemostasis when control of minimal, mild, and moderate bleeding by conventional procedures is ineffective or impractical, except in neurosurgical, ophthalmic, and urological procedures.
  Arms: HEMOBLAST Bellows (Hemostatic Device)
Device: FLOSEAL — The FLOSEAL Matrix consists of a bovine-derived Gelatin Matrix component, a human-derived Thrombin component, applicator tips, and several mixing accessories. FLOSEAL is indicated in surgical procedures (other than ophthalmic) as an adjunct to hemostasis when control of bleeding by ligature or conventional procedures is ineffective or impractical.
  Arms: FLOSEAL (Hemostatic Device)

SUMMARY:
The purpose of this study is to evaluate the performance of HEMOBLAST™ compared to FLOSEAL in cardiothoracic operations.

DETAILED DESCRIPTION:
A maximum of 104 subjects will be enrolled across a maximum of 5 study sites in the United States.

The estimated duration of the study is approximately 8 months from the time of first subject enrollment to the last subject enrollment. Enrollment occurs intraoperatively after confirmation of the intraoperative eligibility criteria. Subjects will undergo intraoperative performance assessments and then will be discontinued from the study after completion of the intraoperative visit.

ELIGIBILITY:
Preoperative Inclusion Criteria

* Subject is undergoing a non-emergent cardiothoracic surgery; and
* Subject or an authorized legal representative is willing and able to give prior written informed consent for study participation.

Preoperative Exclusion Criteria

* Subject has a known sensitivity or allergy to bovine and/or porcine substance(s) or any other component(s) of the hemostatic agent;
* Subject has religious or other objections to porcine or bovine components; and
* Subject is not appropriate for inclusion in the clinical study, per the medical opinion of the Investigator.

Intraoperative Inclusion Criteria

* Subject does not have an active or suspected infection at the surgical site;
* Subject in whom the Investigator is able to identify a Target Bleeding Site (TBS) for which any applicable conventional means for hemostasis are ineffective or impractical; and
* Subject has a TBS with minimal, mild, or moderate bleeding

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Bruckner, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (4):
- United States (4):
  - University of California Los Angeles, Los Angeles, California
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Houston Methodist, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dang NC, Ardehali A, Bruckner BA, Parrino PE, Gillen DL, Hoffman RW, Spotnitz R, Cavoores S, Shorn IJ, Manson RJ, Spotnitz WD. Prospective, multicenter, randomized, controlled trial evaluating the performance of a novel combination powder vs hemostatic matrix in cardiothoracic operations. J Card Surg. 2020 Feb;35(2):313-319. doi: 10.1111/jocs.14376. Epub 2019 Nov 25. PMID 31763732

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One additional subject was enrolled due to a delay in the reporting function of the electronic database used for the study. This additional subject is not anticipated to affect the analyses or ethical conduct of the study, as all subjects were treated on-label for an approved device in this post-market study
Period: Overall Study
Arm/Group | HEMOBLAST Bellows (Hemostatic Device) | FLOSEAL (Hemostatic Device)
Started (1 additional subject enrolled due to delay in reporting function of electronic database.) | 53 | 52
Completed | 53 | 52
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HEMOBLAST Bellows (Hemostatic Device) | FLOSEAL (Hemostatic Device) | Total
Number analyzed (Participants) | 53 | 52 | 105
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.6 (11.4) | 64.9 (12.1) | 63.7 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 8 | 24
  Male | 37 | 44 | 81
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 2 | 10
  Not Hispanic or Latino | 44 | 50 | 94
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 9 | 15 | 24
  Native Hawaiian or Other Pacific Islander | 7 | 6 | 13
  Black or African American | 4 | 6 | 10
  White | 27 | 22 | 49
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: 3 Minute Hemostasis - Hemostatic Success (Yes/no) at 3 Minutes
Description: The primary endpoint of this study is the superiority of HEMOBLAST™ relative to FLOSEAL for the proportion of subjects reaching hemostasis within 3 minutes.
Time Frame: Intraoperative
Measure: Count of Participants; unit: Participants
Arm/Group | HEMOBLAST Bellows (Hemostatic Device) | FLOSEAL (Hemostatic Device)
Number analyzed (Participants) | 53 | 52
Participants | 34 | 5

2. Secondary Outcome: 5 Minute Hemostasis - Hemostatic Success (Yes/no) at 5 Minutes
Description: The secondary endpoint of this study is non-inferiority of HEMOBLAST™ relative to FLOSEAL for the proportion of subjects reaching hemostasis within 5 minutes.
Time Frame: Intraoperative
Measure: Count of Participants; unit: Participants
Arm/Group | HEMOBLAST Bellows (Hemostatic Device) | FLOSEAL (Hemostatic Device)
Number analyzed (Participants) | 53 | 52
Participants | 49 | 23

ADVERSE EVENTS:
Time Frame: Enrollment to discontinuation (intraoperative period, approximately 8 hours))
Description: The rate of occurrence of device malfunctions, device-related adverse events (AEs), serious adverse device effects (SADEs), and unanticipated adverse device effects (UADEs) were summarized for each treatment group by severity.
Arm/Group | HEMOBLAST Bellows (Hemostatic Device) | FLOSEAL (Hemostatic Device)
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/52
Other Adverse Events (participants affected / at risk) | 0/53 | 0/52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-15): https://cdn.clinicaltrials.gov/large-docs/98/NCT03725098/Prot_SAP_000.pdf